CLINICAL TRIAL: NCT02119754
Title: Open Label Trial of Topical PluroGel PN for the Treatment of Patients With Mildly Infected Diabetic Foot Ulcer CLINICAL PROTOCOL PGN-1300X
Brief Title: Topical PluroGel PN for the Treatment of Mildly Infected Diabetic Foot Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PluroGen Therapeutics, Inc (Industry)
Collaborators: Arkios BioDevelopment International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGN-1300X; D11AC00020 (Other Grant/Funding Number: DoD)
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Diabetic Foot Ulcer; Infection
Keywords: Wound; Ulcer; Infected; Infection
MeSH Terms: conditions — Diabetic Foot; Infections; Wounds and Injuries; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plurogel PN (Experimental): Plurogel PN
  Interventions: Drug: Plurogel PN

INTERVENTIONS:
Drug: Plurogel PN

SUMMARY:
This is an open label study of subjects who have failed Protocol PGN-1300. Adult subjects (greater than 18 years old) who present with a mildly infected diabetic foot ulcer (IDSA criteria) having full thickness (i.e., through the dermis but not involving joint capsule, tendon, and bone) and have failed PGN-1300. Subjects must also provide informed consent and meet all other entry criteria to be enrolled and receive PluroGel PN.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have failed treatment on Protocol PGN-1300X

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Clinical Response | 14 days
  Clinical Response is defined by the investigator's evaluation of the signs and symptoms of clinical infection.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Ledesma Foot and Ankle, Phoenix, Arizona
  - Foot & Ankle Clinic, Los Angeles, California
  - Samuel Merritt University, Oakland, California
  - ASAP Urgent-Care, Hamden, Connecticut
  - Advance Medical Research Center, Miami, Florida
  - Miami Center for Clinical Research, LLC, Miami, Florida
  - Unlimited Medical Research, LLC, Miami, Florida
  - Phoenix Medical Research, LLC, Miami, Florida
  - Med Research of Florida, LCC, Miami, Florida
  - Sweet Hope Research Specialty, Inc., Miami Lakes, Florida
  - Weil Foot & Ankle Institute, Des Plaines, Illinois
  - Research Integrity, Owensboro, Kentucky
  - Paddington Testing Company, Inc, Philadelphia, Pennsylvania
  - AllCare Foot & Ankle, PA, Arlington, Texas
  - Coastal Podiatry Group, Virginia Beach, Virginia